CLINICAL TRIAL: NCT06408688
Title: Safety and Modulation of Adaptive Immunity by Iscador® Qu Viscum Album Extract in Patients With Advanced, Recurrent or Metastatic Cancers Treated With Immune Checkpoint Inhibitors - a Randomized Trial
Brief Title: Safety and Modulation of Adaptive Immunity by Iscador® Qu Viscum Album Extract in Patients With Advanced, Recurrent or Metastatic Cancers Treated With Immune Checkpoint Inhibitors
Acronym: ISCA-CHECK
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-02373; th23binder
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Advanced Solid Tumor
Keywords: Mistletoe Extract
MeSH Terms: interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Immune checkpoint inhibitors plus Iscador® Qu (Active Comparator): Patients randomized to Arm A will be treated with Immune checkpoint inhibitors plus Iscador® Qu.
  Interventions: Drug: Immune checkpoint inhibitors plus Iscador® Qu.
- Arm B: Immune checkpoint inhibitors (Active Comparator): Patients randomized to Arm B will be treated with Immune checkpoint inhibitors only.
  Interventions: Drug: Immune Checkpoint Inhibitors

INTERVENTIONS:
Drug: Immune checkpoint inhibitors plus Iscador® Qu. — Standard cancer treatment plus subcutaneous injection of mistletoe fermented extract (Iscador® Qu) as per the summary of product characteristics.
  Arms: Arm A: Immune checkpoint inhibitors plus Iscador® Qu
Drug: Immune Checkpoint Inhibitors — Standard cancer treatment.
  Arms: Arm B: Immune checkpoint inhibitors

SUMMARY:
The main objective of this study is to test if adding the mistletoe extract Iscador® Qu to regular cancer treatment with immune checkpoint inhibitors affects:

* The immune system's ability to fight cancer
* Safety of the treatment
* How well the treatment performs against cancer
* How the patient feels during treatment

Researchers will compare patients treated with immune checkpoint inhibitors plus Iscador® Qu with patients treated with imune checkpoint inhibitors only.

DETAILED DESCRIPTION:
The impact of mistletoe preparations - that are claimed to have immunostimulatory properties - on cancer treatment with immune checkpoint inhibitors remains unclear. To address this knowledge gap, the current study aims to investigate the modulation of adaptive immunity through the combination of Iscador (a specific mistletoe preparation) and immune checkpoint inhibitors. Additionally, researchers will evaluate the safety profile of this combination therapy in patients with locally advanced non-operable or metastatic cancers except for skin cancers. By examining the modulation of adaptive immunity and safety of this treatment approach, researchers aim to provide valuable insights for clinicians and patients in the context of advanced cancer care.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced non-operable or metastatic solid tumor, except for skin cancer
* Eligible for routine (standard) treatment with immune checkpoint inhibitor (+/- chemo/targeted therapy) as per the discretion of the local investigator
* Subjects must be eligible for treatment with mistletoe preparations (controlled brain metastases, prednisolone equivalent below 10mg, no known hypersensitivity)
* ECOG (Eastern Cooperative Oncology Group) performance status score of 0-2
* Males and Females at least 18 years of age; no subjects under tutelage
* No previous mistletoe treatment

Exclusion Criteria:

* Contraindications to Iscador® Qu or immune checkpoint inhibitors, e.g. hypersensitivity, active autoimmune disorder
* Patients with skin cancer
* Participation in another study with investigational drug within 30 days prior to enrolment (participation in observational studies or diagnostic studies without a particular drug intervention are allowed)
* Enrolment of the investigator, his/her family members, employees and other dependent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with a relative increase in T cell richness or diversity of 20% or more | baseline and 12 weeks (+/- 2 weeks)
  Percentage of patients with a relative increase in T cell richness or diversity of 20% or more as measured by peripheral blood T cell receptor Next-generation sequencing.
Percentage of patients with a relative decrease in T cell clonality of 20% or more | baseline and 12 weeks (+/- 2 weeks)
  Percentage of patients with a relative decrease in T cell clonality of 20% or more as measured by peripheral blood T cell receptor Next-generation sequencing.
Level of T cell richness | baseline and 12 weeks (+/- 2 weeks)
  Level of T cell richness as measured by peripheral blood T cell receptor Next-generation sequencing.
Level of T cell diversity | baseline and 12 weeks (+/- 2 weeks)
  Level of T cell diversity as measured by peripheral blood T cell receptor Next-generation sequencing.
Level of T cell clonality | baseline and 12 weeks (+/- 2 weeks)
  Level of T cell clonality as measured by peripheral blood T cell receptor Next-generation sequencing.

SECONDARY OUTCOMES:
Safety and tolerability according to the NCI CTC AE v5 | up to 18 weeks
  Safety and tolerability according to the NCI CTC AE v5 (National Cancer Institute Common Terminology Criteria for Adverse Events)
Rate of early immune checkpoint inhibitor-based treatment termination | up to 24 months
  Rate of early immune checkpoint inhibitor-based treatment termination
Best tumor response | up to 24 months
  Best tumor response as per investigators assessment
Progression-free survival | up to 24 months
  Investigator-assessed progression-free survival
Overall survival | up to 24 months
  Overall survival
EORTC QLQ C30 | up to 24 months
  Quality of life as measured by EORTC QLQ C30 (European Organisation for Research and Treatment of Cancer, Quality of Life Questionnaire). Calculation of the scores follows the validated formulas as issued by the EORTC. Scores range from 0% to 100% for all questionnaire domains with higher values representing better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Kasenda, PD Dr. Dr., Principal Investigator — USB
Locations (4):
- Switzerland (4):
  - Kantosspital Baden AG, Baden
  - Universitätsspital Basel, Basel
  - Kantonsspital Baselland, Liestal
  - Tumor- und Brustzentrum Ostschweiz, Sankt Gallen

IPD SHARING:
Plan to Share IPD: No